CLINICAL TRIAL: NCT01145508
Title: Randomized Phase II Trial of Docetaxel With or Without PSA-TRICOM Vaccine in Patients With Castrate-Resistant Metastatic Prostate Cancer
Brief Title: Docetaxel and Prednisone With or Without Vaccine Therapy in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02048; NCI-2011-02048 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000675173; E1809; E1809 (Other: ECOG-ACRIN Cancer Research Group); E1809 (Other: CTEP); U10CA180820 (NIH); U10CA021115 (NIH)
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Hormone-Resistant Prostate Cancer; Prostate Adenocarcinoma; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone; deltacortene; prednylidene; PROSTVAC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (vaccine therapy and chemotherapy) (Experimental): Patients receive rilimogene-galvacirepvec SC on day 1 of course 1 and fowlpox-PSA-TRICOM vaccine SC on days 15, 29, 43, and 57 of course 1. Beginning on day 85 (day 1 of course 2), patients receive docetaxel IV over 1 hour on day 1 and prednisone PO BID on days 1-21. Treatment with docetaxel and prednisone repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Drug: Prednisone; Biological: Recombinant Fowlpox-PSA(L155)/TRICOM Vaccine; Biological: Rilimogene Galvacirepvec
- Arm B (docetaxel, prednisone) (Active Comparator): Patients receive docetaxel IV over 1 hour on day 1 and prednisone PO BID on days 1-21. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Drug: Prednisone

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Biological: Recombinant Fowlpox-PSA(L155)/TRICOM Vaccine — Given SC
  Other Names: PROSTVAC-F; rFowlpox-PSA(L155)/TRICOM Vaccine
  Arms: Arm A (vaccine therapy and chemotherapy)
Biological: Rilimogene Galvacirepvec — Given SC
  Other Names: PROSTVAC; Prostvac-V; Recombinant Vaccinia-PSA(L155)-TRICOM Vaccine; Recombinant Vaccinia-PSA(L155)/TRICOM; Recombinant Vaccinia-PSA(L155)/TRICOM Vaccine; rVaccinia-Prostate-Specific Antigen/TRICOM Vaccine; rVaccinia-PSA(L155)-TRICOM Vaccine
  Arms: Arm A (vaccine therapy and chemotherapy)

SUMMARY:
This randomized phase II trial studies how well docetaxel and prednisone with or without vaccine therapy works in treating patients with hormone-resistant prostate cancer that has spread to other parts of the body. Drugs used in chemotherapy, such as docetaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Vaccines made from an antigen may help the body build an effective immune response to kill tumor cells. It is not yet known whether docetaxel and prednisone are more effective with or without vaccine therapy in treating prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the overall survival in patients treated with PSA-TRICOM (fowlpox-PSA-TRICOM vaccine and rilimogene-galvacirepvec) and docetaxel chemotherapy versus docetaxel chemotherapy only.

SECONDARY OBJECTIVES:

I. To evaluate the time to radiographic progression after beginning docetaxel chemotherapy in patients previously treated with PSA-TRICOM vaccine versus those not treated with this vaccine.

II. To compare objective responses (according to Response Evaluation Criteria in Solid Tumors [RECIST]) between the two treatment groups in those patients with measurable disease.

III. To evaluate prostate-specific antigen (PSA) response rates (decline >= 50%) in patients treated with PSA-TRICOM and docetaxel chemotherapy versus docetaxel chemotherapy only.

IV. To evaluate immune responses elicited in patients treated before and after docetaxel chemotherapy.

V. To evaluate the association between development of prostate antigen-specific immune responses and time to progression and overall survival.

VI. To evaluate the association of predicted survival (by Halabi nomogram) with actual survival in patients treated with PSA-TRICOM vaccine versus those not treated with this vaccine.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A (vaccine and chemotherapy): Patients receive rilimogene-galvacirepvec subcutaneously (SC) on day 1 of course 1 and fowlpox-PSA-TRICOM vaccine SC on days 15, 29, 43, and 57 of course 1. Beginning on day 85 (day 1 of course 2), patients receive docetaxel intravenously (IV) over 1 hour on day 1 and prednisone orally (PO) twice daily (BID) on days 1-21. Treatment with docetaxel and prednisone repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

ARM B (chemotherapy): Patients receive docetaxel IV over 1 hour on day 1 and prednisone PO BID on days 1-21. Treatment repeats every 21 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically confirmed diagnosis of prostate cancer (adenocarcinoma of the prostate)
* Patient must have metastatic disease as evidenced by the presence of soft tissue and/or bone metastases on imaging studies (computed tomography [CT] of abdomen/pelvis, bone scintigraphy)
* Patient must have castrate-resistant disease, defined as follows:

  * Patient must have received standard of care androgen deprivation treatment (ADT) before trial entry (surgical castration versus gonadotropin-releasing hormone [GnRH] analogue or antagonist treatment); subjects receiving GnRH analogue or antagonist must continue this treatment throughout the time on this study
  * Patient must have been treated previously with a nonsteroidal antiandrogen, with evidence of subsequent disease progression; subjects must be off use of anti-androgen for at least 4 weeks (for flutamide) or 6 weeks (for bicalutamide or nilutamide) prior to randomization; subjects who demonstrate an anti-androgen withdrawal response, defined as a >= 25% decline in PSA within 4-6 week of stopping a nonsteroidal antiandrogen are not eligible until the PSA rises above the nadir observed after antiandrogen withdrawal
  * Patient must have castration levels of testosterone (< 50 ng/dL) within 4 weeks prior to randomization
* Patient must have progressive disease while receiving ADT as defined by any one of the following as per the Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria:

  * PSA: at least two consecutive rises in serum PSA, obtained at a minimum of 1-week intervals, and each value >= 2.0 ng/mL
  * Measurable disease: >= 50% increase in the sum of the cross products of all measurable lesions or the development of new measurable lesions by RECIST criteria version 1.1; the greatest diameter of a target lesion must be at least 1.0 cm by CT scan (1.5 cm in shortest axis for lymph nodes)
  * Non-measurable (bone) disease: the appearance of two or more new areas of uptake on bone scan consistent with metastatic disease compared to previous imaging during castration therapy; the increased uptake of pre-existing lesions on bone scan will not be taken to constitute progression, and ambiguous results must be confirmed by other imaging modalities (e.g. X-ray, CT or magnetic resonance imaging [MRI])
* Patient must not have poor prognosis features suggested by the following required information:

  * Presence of visceral (non-lymph node, non-bone) metastases
  * Poor performance status (Eastern Cooperative Oncology Group [ECOG] performance status [PS] of 2 or greater)
  * Alkaline phosphatase (IU/L) > 2 x institutional upper limit of normal
  * Lactate dehydrogenase (LDH) (U/L) > 2 x institutional upper limit of normal
* Patient must have an ECOG performance status of 0 or 1
* White blood cell (WBC) count >= 2000/mm^3
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine =< 2.0 mg/dL
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) =< 1.5 x institutional upper limit of normal (ULN)
* Total bilirubin < institutional upper limit of normal (ULN)
* Patient must have completed any prior treatments (apart from androgen deprivation as previously described) >= 4 weeks prior to randomization and have recovered (to < grade 2) from any acute toxicities attributed to this prior treatment
* Patient must agree to use an accepted and effective method of contraception prior to study entry and for the duration of study participation (or at least 4 months after the last vaccination in subjects receiving vaccine series); if patient impregnates a woman while participating in this study, he should inform his treating physician immediately
* Patient must not be receiving any other investigational agents or be receiving concurrent anticancer therapy other than ADT
* Patient must not have been treated with a prior anti-cancer vaccine (including sipuleucel-T, Provenge®)
* Patient must not have received treatment with any of the following medications within 4 weeks of randomization or while on study:

  * Systemic corticosteroids (excluding prednisone and dexamethasone administered as part of study protocol); inhaled, intranasal or topical corticosteroids are acceptable; steroid eye drops are contraindicated however, for 2 weeks prior to vaccination and for at least 4 weeks after vaccinia vaccination
  * PC-SPES
  * Saw palmetto
  * Megestrol
  * Ketoconazole
  * 5-alpha-reductase inhibitors - patients already taking 5-alpha-reductase inhibitors prior to 28 days prior to randomization may stay on these agents throughout the course of therapy, but these should not be started while patients are on study
  * Diethyl stilbestrol
  * Any other hormonal agent or supplement with possible anti-cancer activity
* Patient must not have been treated with external beam radiation therapy within 4 weeks of randomization
* Patient must not have received prior radiation therapy to > 30% of bone marrow
* Patient must not have had surgery within 4 weeks of randomization
* Patient must not have received prior chemotherapy within 6 months of randomization; prior and/or concurrent treatment with bisphosphonates, however, is permitted
* Patient must not have received prior chemotherapy for metastatic prostate cancer
* Patient cannot have a known history of human immunodeficiency virus (HIV) 1 or 2, human T-lymphotropic virus (HTLV)-1, hepatitis B, or hepatitis C (or any other potentially immunosuppressive infection); eligible subjects must have negative serologic testing for HIV, hepatitis B surface antigen, and hepatitis C
* Patient cannot have a history of autoimmune disease requiring active immunosuppressive therapy or have organ dysfunction >= grade 2 as a result of known autoimmune disease; eligible subjects must have antinuclear antibodies (ANA) titer < 1:320
* Patient must not have undergone splenectomy
* Patient must not have other active malignancies other than non-melanoma skin cancers or carcinoma in situ of the bladder; subjects with a history of other cancers who have been adequately treated and have been recurrence-free for >= 3 years are eligible
* Patient cannot have a known allergy to eggs
* Patient cannot have a known intolerance or allergic reactions to docetaxel or compounds of similar chemical or biologic composition
* Patient cannot have a known history of allergy or intolerable reaction to a previous vaccinia virus vaccination (e.g., smallpox)
* Patient or close household contacts of patient (those who share housing or have close physical contact with the patient) cannot have close physical contact to persons with the following conditions within 3 weeks after potential vaccinia immunization:

  * A history of eczema, active eczema or other acute, chronic or exfoliative skin conditions, including Darier's disease (e.g. atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or open wounds)
  * Pregnant or nursing women
  * Children under 3 years of age
  * Immunodeficient or immunosuppressed persons (e.g. HIV, or treated for other diseases with immunosuppressive agents)
  * Any other moderate or severe acute illness until the illness resolves Patients who would be unable to avoid these conditions for a 3-week period are not eligible; patients should also refer to the patient instruction sheet for vaccinia virus
* Patient cannot have known brain metastases
* Patient cannot have a known history of recent (within 6 months) stroke, myocardial infarction, unstable angina, New York Heart Association class II-IV congestive heart failure, or significant cardiomyopathy requiring treatment
* Patient cannot take known strong inducers or inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) within 2 weeks of beginning docetaxel through its discontinuation; substrates of CYP3A4 with a narrow therapeutic/toxicity window may be used with caution, with prior approval of the study chair or institution's principal investigator (PI)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2012-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McNeel, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (14):
- United States (14):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - NorthShore Hematology Oncology-Libertyville, Libertyville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Eastern Cooperative Oncology Group (ECOG) member institutions between December 29, 2010 and March 26, 2012.
Groups:
- Arm A (Vaccine and Chemotherapy): Patients receive vaccinia-PSA(L155)-TRICOM vaccine subcutaneously (SC) on day 1 and fowlpox-PSA(L155)-TRICOM vaccine SC on days 15, 29, 43, and 57. Beginning on day 85, patients receive chemotherapy in a 21-day cycle. Docetaxel is administered intravenously (IV) over 1 hour on day 1. Prednisone is given orally (PO) twice daily on days 1-21. Treatment with docetaxel and prednisone repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  PSA-TRICOM vaccine: Given SC
  fowlpox-PSA-TRICOM vaccine: Given SC
  docetaxel: Given IV
  prednisone: Given PO
- Arm B (Chemotherapy): Patients receive docetaxel IV over 1 hour on day 1 and prednisone PO twice daily on days 1-21. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  docetaxel: Given IV
  prednisone: Given PO
Period: Overall Study
Arm/Group | Arm A (Vaccine and Chemotherapy) | Arm B (Chemotherapy)
Started | 7 | 3
Treated | 6 | 2
Completed | 2 | 1
Not Completed | 5 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Never started treatment | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Vaccine and Chemotherapy) | Arm B (Chemotherapy) | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Continuous [Median (Full Range); unit: years] | 63 [56 to 72] | 65 [65 to 73] | 64 [56 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to death or the date of last known alive.
Time Frame: Assessed every 3 months for 2 years, and then every 6 months for 3 years
Population: All randomized patients are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Vaccine and Chemotherapy) | Arm B (Chemotherapy)
Number analyzed (Participants) | 7 | 3
Months | 20.8 [3.4 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [14.8 to NA] — The median was not reached and the upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Arm/Group | Arm A (Vaccine and Chemotherapy) | Arm B (Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 5/6 | 2/2
Other Adverse Events (participants affected / at risk) | 5/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Vaccine and Chemotherapy) (N=6) | Arm B (Chemotherapy) (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 4 | 2
White blood cell decreased (Investigations) | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Vaccine and Chemotherapy) (N=6) | Arm B (Chemotherapy) (N=2)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Chills (General disorders) | 1 | 0
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 3 | 1
Fatigue (General disorders) | 5 | 2
Fever (General disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue - Other (Skin and subcutaneous tissue disorders) | 2 | 1
Bloating (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Creatinine increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 3 | 2
Headache (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 1
Watering eyes (Eye disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less